CLINICAL TRIAL: NCT01847482
Title: COOL-ARREST JP: A Multicenter, Prospective, Single-arm Interventional Trial to Evaluate Therapeutic Hypothermia With IntraVascular Temperature Management (IVTM) in Post-Cardiogenic Cardiac Arrest and Post-Return of Spontaneous Circulation Patients
Brief Title: Therapeutic Hypothermia With IntraVascular Temperature Management (IVTM) in Post-Cardiogenic Cardiac Arrest and Post-Return of Spontaneous Circulation Patients in Japan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ZOLL Circulation, Inc., USA (Industry)
Collaborators: Asahi Kasei Medical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COOL-ARREST JP
Record Dates: First submitted 2013-02-11; First posted 2013-05-06 (Estimated); Last update posted 2018-06-27 (Actual); Status verified 2014-06

CONDITIONS: Cardiac Arrest
Keywords: Cardiac arrest; Return of Spontaneous Circulation (ROSC); IntraVascular Temperature Management (IVTM); Therapeutic Hypothermia; Japan
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Therapeutic Hypothermia (Experimental)
  Interventions: Device: ZOLL Intravascular Temperature Management System (IVTM)

INTERVENTIONS:
Device: ZOLL Intravascular Temperature Management System (IVTM) — Induced therapeutic hypothermia post cardiac arrest

SUMMARY:
A multicenter, single-arm, prospective, interventional trial to evaluate therapeutic hypothermia with intravascular temperature management (IVTM) in post-cardiogenic cardiac arrest, post-return of spontaneous circulation (ROSC) patients in Japan.

The objective of this study is to verify that therapeutic hypothermia performed by intravascular cooling using the investigational device (IVTM) can control body temperature appropriately in post-cardiogenic cardiac arrest, post-ROSC patients.

ELIGIBILITY:
Inclusion Criteria:

1. Non-traumatic in-hospital or out-of-hospital cardiac arrest
2. Unwitnessed cardiac arrest (Ventricular fibrillation), or witnessed cardiac arrest (ventricular fibrillation, pulseless electrical activity, asystole within 15 minutes following onset)
3. Patient is at least 20 years of age and less than 80 years of age with consent is given
4. In the judgement of an investigator or sub-investigator, the patient is unable to follow verbal instructions
5. Therapeutic hypothermia using the investigational device can be initiated within six hours of Return of Spontaneous Circulation (ROSC)
6. Written consent can be obtained from a legally acceptable representative

Exclusion Criteria:

1. Traumatic cardiac arrest (blunt trauma, penetrating trauma, burns, exsanguination, suffocation, smoke inhalation, near drowning, etc)
2. Accidental hypothermia with core body temperature less than 35.0°C
3. Pregnant or of child bearing potential
4. Patient has given or indicated a Do Not Resuscitate (DNR) order
5. Femoral venous access is contraindicated by previous surgey, medical history, anatomy or the like
6. An inferior vena cava filter is in place
7. Patient has severe bleeding (Pulmonary hemorrhage, gastrointestinal hemorrhage, etc.)
8. Intracranial hemorrhage as confirmed by CT scanning
9. Hemodynamic instability despite use of vasopressor agents and cardiac stimulants
10. Heparin hypersensitivity
11. Serious systemic infectious diseases (sepsis, etc.)
12. Platelet count less than 30,000/mm3
13. Serious hepatic dysfunction
14. Serious renal impairment
15. Using percutaneous cardiopulmonary support (PCPS)
16. Using continuous hemodiafiltration (CHDF)
17. Therapeutic hypothermia has been otherwise implemented between ROSC and the start of the study (excluding the rapid infusion of non-glucose-containing cold electrolyte fluid, or non-glucose-containing cold plasma volume expander)
18. The patient's core body temperature cannot be monitored
19. Currently participating in another clinical trial or has participated in another clinical trial within the past six months
20. in the judgement of an investigator or sub-investigator, participation in this clinical trial is inappropriate for the patient

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2013-03; Primary Completion 2014-06 (Actual); Study Completion 2016-01-19 (Actual)

PRIMARY OUTCOMES:
Core temperature achievement ratio | Baseline and 3 hours

SECONDARY OUTCOMES:
Cerebral Performance Category (CPC) | Baseline and 14 days
Modified Rankin Scale (mRS) | Baseline and 14 days
Change in body temperature | Baseline and 96 hours
Cooling speed | Baseline and 3 hours
Safety | Baseline vs. 2 days
  Incidence of adverse events at 2 days compared to baseline.
Safety | Baseline vs. 14 days
  Incidence of adverse events at 14 days compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Yoichi Kato, PhD, Study Director — Asahi Kasei Medical Co., Ltd.; Tsuyoshi Maekawa, MD, PhD, Principal Investigator — Yamaguchi Grand Medical Center
Locations (10):
- Japan (10):
  - Kokura Memorial Hospital, Kitakyushu, Fukuoka
  - Sapporo Medical University Hospital, Sapporo, Hokkaido
  - Hyogo College of Medicine Hospital, Nishinomiya, Hyōgo
  - Iwate Medical University Hospital, Morioka, Iwate
  - Kagawa University School of Medicine, Hiragi, Kagawa-ken
  - Nipponn Medical School Hospital, Bunkyo, Tokyo
  - Surugadai Nihon University Hospital, Chiyoda City, Tokyo
  - Yamaguchi University Hospital, Ube, Yamaguchi
  - National Hospital Organization Kumamoto Medical Center, Kumamoto
  - Osaka City General Hospital, Osaka